CLINICAL TRIAL: NCT02318095
Title: Feasibility Study of Neoadjuvant Gemcitabine/Nab-Paclitaxel and Hypofractionated Image-Guided Intensity Modulated Radiotherapy in Resectable and Borderline Resectable Pancreatic Cancer
Brief Title: Gemcitabine/Nab-Paclitaxel With HIGRT in Resectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00058865
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Resectable Pancreatic Cancers
Keywords: Cancer of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy/radiation/surgery (Other): This is a single arm prospective study. All eligible subjects will recieve 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel, followed by hypofractionated radiation therapy followed by surgical resection. Subjects may receive adjuvant chemotherapy post surgical resection at the clinical discretion of the medical oncologist.
  Interventions: Drug: Gemcitabine/nab-Paclitaxel; Radiation: Radiation therapy; Other: Sugical resection; Drug: Adjuvant chemotheapy

INTERVENTIONS:
Drug: Gemcitabine/nab-Paclitaxel — Prospective, single arm study ; eligible subjects will recieve 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel. All chemotherapy administered to study subjects is standard of care. The chemotherapy combination, gemcitabine/nab-paclitaxel, is considered to be a standard-of-care, non-investigational chemotherapy combination; chemotherapy dosing and treatment schedule will be managed by the treating medical oncologist. Restaging will be completed post chemotherapy.
Radiation: Radiation therapy — 5 fractions of hypofractionated IGRT or IMRT at 5Gy per fraction will be delivered before surgery. Restaging will be completed post radiation therapy.
Other: Sugical resection — Surgical resection of the pancreas post radiation therapy
Drug: Adjuvant chemotheapy — Adjuvant chemotherapy may be given after surgery at the clinical discretion of the medical oncologist

SUMMARY:
This research protocol will evaluate the feasibility of administering neoadjuvant gemcitabine and nab-paclitaxel with hypofractionated, image guided, intensity modulated radiotherapy (HIGRT) in resectable and borderline resectable pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer-related death in the United States and accounts for roughly 40,000 deaths each year. Despite the use of neoadjuvant and adjuvant therapies, little progress has been made in the the last three decades, and the search for more efficacious treatment continues.In patients with a good performance status the combination of effective systemic therapy with gemcitabine/nab-paclitaxel and high dose local radiotherapy may improve disease outcomes. This is a prospective, single arm study in patients in newly diagnosed, previously untreated pancreatic cancer who are planned to undergo surgical resection The primary objective of this study is to evaluate the toxicity of a neoadjuvant approach incorporating gemcitabine/nab-paclitaxel and Hypofractionated image guided intensity-modulated radiotherapy (HIGRT) prior to surgical resection. Eligible subjects will recieve standard neoadjuvant gemcitabine and nab-paclitaxel dosing is as follows:Nab-Paclitaxel (125mg/m2) days 1,8,15 every 28 days for 2 cycles Gemcitabine (1000mg/m2) days 1,8,15 every 28 days for 2 cycles followed by HIGRT and surgical resection.

Adjuvant chemotherapy may be given post surgery at the discretion of the treating medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed informed consent and is willing to comply with the protocol
2. Histologically or cytologically proven adenocarcinoma of the pancreas (within the last 90 days)
3. Either resectable or borderline resectable as determined on staging imaging (as defined by National Comprehensive Cancer Network [NCCN])
4. Patient is 18 years or older
5. Karnofsky performance status 70 or greater
6. The ANC count ≥ 1500, the platelet count ≥ 100,000 and hemoglobin ≥ 9g/dL
7. Laboratory values meet the following constraints: Bilirubin less than or equal to 2 mg/dL; AST and ALT less than or equal to 3 x ULN (stenting to improve biliary obstruction is permitted)
8. No evidence of metastatic disease based on imaging of the chest, abdomen and pelvis.

Exclusion Criteria:

1. Metastatic disease on pretreatment imaging
2. Prior systemic therapy
3. Prior abdominal radiation. Any prior radiation must be approved by the Radiation Oncology PI
4. Previous treatment for pancreatic cancer
5. Patients with any serious/poorly controlled medical or psychological conditions that would be exacerbated by treatment, would complicate protocol compliance
6. Pregnant or lactating. Adequate birth control must be used if of child bearing potential per institutional policy. Negative pregnancy test in female patients of child-bearing potential per institutional policy. Post-menopausal women must have had amenorrhea for at least 18 months to be considered non-child bearing
7. Clinically significant peripheral vascular disease
8. Presence of active or chronic infection
9. Clinically significant atherosclerotic cardiovascular disease including patients with New York Heart Class II/III/IV CHF, ventricular arrhythmias requiring medication, myocardial infarction, cerebrovascular accident, transient ischemic attack, coronary artery bypass grafting, angioplasty, cardiac or other vascular stenting within the past 6 months
10. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess within six months prior to treatment start
11. History of collagen vascular disease or inflammatory bowel disease (Crohn's or ulcerative colitis)
12. Current grade 2 or higher peripheral neuropathy
13. Anticoagulation with warfarin
14. History of arterial thromboembolic events or symptomatic pulmonary embolism within the past 6 months
15. Active bleeding diathesis or history of major bleeding, CNS bleeding, or significant hemoptysis within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy/Radiation/Surgery: This is a single arm prospective study. All eligible subjects will receive 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel, followed by hypofractionated radiation therapy followed by surgical resection. Subjects may receive adjuvant chemotherapy post surgical resection at the clinical discretion of the medical oncologist.
  Radiation therapy: 5 fractions of hypofractionated IGRT or IMRT at 5Gy per fraction will be delivered before surgery. Restaging will be completed post radiation therap
Period: Overall Study
Arm/Group | Chemotherapy/Radiation/Surgery
Started | 40
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy/Radiation/Surgery: Gemcitabine/nab-Paclitaxel: Prospective, single arm study ; eligible subjects will recieve 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel. All chemotherapy administered to study subjects is standard of care. The chemotherapy combination, gemcitabine/nab-paclitaxel, is considered to be a standard-of-care, non-investigational chemotherapy combination; chemotherapy dosing and treatment schedule will be managed by the treating medical oncologist. Restaging will be completed post chemotherapy.
  Radiation therapy: 5 fractions of hypofractionated IGRT or IMRT at 5Gy per fraction will be delivered before surgery. Restaging will be completed post radiation therap
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Participants Who Complete the Neoadjuvant Gemcitabine/Nab-paclitaxel and HIGRT Regimen
Description: The neoadjuvant regimen will be considered feasible if (a) the trial can accrue 25 patients in no more than 3 years and (b) if at least 17 of the 25 patients adhere to the neoadjuvant regimen and c) the acute grade 3+ non-hematologic acute toxicity is less than 50% (exclusing fatigue and alopecia).
Time Frame: approximately 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Chemotherapy/Radiation/Surgery: This is a single arm prospective study. All eligible subjects will receive 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel, followed by hypofractionated radiation therapy followed by surgical resection. Subjects may receive adjuvant chemotherapy post surgical resection at the clinical discretion of the medical oncologist.
  Radiation therapy: 5 fractions of hypofractionated IGRT or IMRT at 5Gy per fraction will be delivered before surgery. Restaging will be completed post radiation therapy.
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 40
Participants | 39

2. Secondary Outcome: Number of Participants Experiencing Grade >/=2 Acute Toxicity
Description: CTCAE version 4 will be used for all toxicity assessments. The acute toxicity rate, defined as any non-hematologic grade 2+ toxicity occurring during HIGRT treatment through 60 days post-treatment, will be estimated with its exact 80% confidence interval. Likewise, we will determine the rate of grade 2+ hematologic toxicity occurring during treatment through 60 days post treatment and the proportion of patients requiring treatment breaks longer than 5 days.
Time Frame: 60 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 40
Participants | 10

3. Secondary Outcome: Number of Participants Who Underwent Surgical Resection
Description: Patients who undergo surgical resection will be documented
Time Frame: 14-30 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 40
Participants | 24

4. Secondary Outcome: Number of Participants Who Received an R0 Resection
Description: Pathologic review will determine if an R0 resection has been performed. R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Time Frame: 14-30 days post surgery
Population: Participants who underwent surgical resection.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy/Radiation/Surgery
Number analyzed (Participants) | 24
Participants | 18

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of HIGRT through 60 days post surgery, about 6 months.
Groups:
- Chemotherapy/Radiation/Surgery: This is a single arm prospective study. All eligible subjects will recieve 2 cycles of neoadjuvant Gemcitabine/nab-Paclitaxel, followed by hypofractionated radiation therapy followed by surgical resection. Subjects may receive adjuvant chemotherapy post surgical resection at the clinical discretion of the medical oncologist.
  Radiation therapy: 5 fractions of hypofractionated IGRT or IMRT at 5Gy per fraction will be delivered before surgery. Restaging will be completed post radiation therap
Arm/Group | Chemotherapy/Radiation/Surgery
All-Cause Mortality (participants affected / at risk) | 24/40
Serious Adverse Events (participants affected / at risk) | 3/40
Other Adverse Events (participants affected / at risk) | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy/Radiation/Surgery (N=40)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 3 (3)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy/Radiation/Surgery (N=40)
Anemia (Blood and lymphatic system disorders) | 6 (7)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (10)
Bloating (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 16 (17)
Diarrhea (Gastrointestinal disorders) | 17 (19)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 27 (33)
Vomiting (Gastrointestinal disorders) | 11 (14)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 5 (5)
Fatigue (General disorders) | 30 (34)
Fever (General disorders) | 6 (7)
Flu like symptoms (General disorders) | 6 (8)
Pain (General disorders) | 13 (13)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (7)
Wound infection (Infections and infestations) | 4 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (6)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 5 (6)
Neutrophil count decreased (Investigations) | 20 (43)
Platelet count decreased (Investigations) | 13 (22)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 11 (15)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4)
Nervous system disorders (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 (8)
Hematoma (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT02318095/Prot_SAP_000.pdf